CLINICAL TRIAL: NCT01456585
Title: Phase 1 Study of Preoperative Gemcitabine Plus CP-870,893 Followed by Addition of CP-870,893 to Standard -Of-care Adjuvant Chemoradiation for Patient With Newly Diagnosed Resectable Pancreatic Carcinoma
Brief Title: Phase 1 Study of Preoperative Gemcitabine Plus CP-870, 893 Followed by Addition of CP-870,893 to Standard -Of-care Adjuvant Chemoradiation for Patients With Newly Diagnosed Resectable Pancreatic Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 14211
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Adenocarcinoma Pancreas
Keywords: Histological documentation; primary adenocarcinoma of the pancreas; surgically eligible; tumor resection; curative intent
MeSH Terms: interventions — Gemcitabine; selicrelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Gemcitabine
Drug: CP-870,893

SUMMARY:
This is a pilot study to evaluate the role of the addition of CP870, 893 to the neoadjuvant and adjuvant setting for patients with resectable pancreatic cancer. Patients will receive standard surgery followed by chemoradiation for their disease, but one dose of gem/cp 870,893 will be pre-op and 3 doses post-op.

DETAILED DESCRIPTION:
This is an open-label single-arm,phase 1, trial. Ten patients with newly diagnosed resectable pancreatic carcinoma will receive gemcitabine and CP-870,893 two weeks prior to surgical resection and subsequently during standard-of-care adjuvant chemoradiation therapy (at which time CP-870,893 will be given on day 3 of each of three 28-day cycles of gemcitabine). Previously established doses of each agent will be used and each given by IV infusion.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of primary adenocarcinoma of the pancreas
* Surgically eligible for tumor resection with curative intent
* Age> 18 years old
* ECOG PS 0 or 1
* Adequate bone marrow function (WBC>3,000; Hgb>9; Plt>100)
* Adequate renal function (Cr<1.5ULN)
* Adequate hepatic function (total bilirubin WNL unless associated with hepatobiliary metastases or Gilbert syndrome, then total bilirubin <2x ULN; and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN
* Signed, written informed consent

Exclusion Criteria:

* Non ductal adenocarcinomas, neuroendocrine neoplasms, cystic tumors of the pancreas such as cystadenomas, cystadenocarcinomas and solid pseudopapillary neoplasms. In addition adenocarcinomas arising from duodenum, distal bile duct, and ampulla will also be excluded.
* Patients with M1 disease.
* Patients with any type of recurrent pancreatic adenocarcinoma
* Prior therapy such as chemotherapy or radiation therapy for pancreatic cancer
* Patients with a previous history of active malignancy within 5 years prior to study entry, except 1) in situ cervical carcinoma or 2) non-melanoma skin cancer
* Previous treatment with any other compound that targets CD40
* Concurrent treatment with any anticancer agent outside of this protocol.
* Prior allogeneic bone marrow transplant
* History of autoimmune disorder, including type 1 diabetes mellitus, pemphigus vulgaris, systemic mastocytosis, systemic lupus erythromatosis, dermatomyositis/polymyositis, rheumatoid arthritis, systemic sclerosis, Sjorgen's syndrome, vasculitis/arteritis, Behcet's syndrome, autoimmune thyroiditis, multiple sclerosis, or uveitis. Vitiligo is allowed.
* History (within the previous year) of stroke or transient ischemic attack, unstable angina, myocardial infarction, congestive heart failure.
* History of deep venous thrombosis or migratory thrombophlebitis (Trousseau);
* Hereditary or acquired coagulopathies (e.g., hemophilia, von Willebrands's disease, or cancer-associated DIC)
* Prior allergic reactions attributed to other monoclonal antibodies.
* Concurrent or planned concurrent treatment with systemic high dose (immunosuppressive) corticosteroids or treatment with systemic corticosteroids within 4 weeks of baseline.
* Treatment on another therapeutic clinical trial within 4 weeks of enrollment in this trial.
* Concurrent or planned concurrent treatment with anticoagulant such as Coumadin or heparin, except to maintain patency of in-dwelling catheters.
* Ongoing or active infection;treatment with systemic antibiotics or antifungals for ongoing or recurrent infection (topical use of antibiotics or antifungals is allowed)
* Pregnancy or breast-feeding-female patients must be surgically sterile, be post-menopausal, or must agree to use effective contraception during the period of therapy and for 12 months following the last dose of CP-870,893. All female patients with reproductive potential may not participate unless they agree to use an effective contraceptive method.
* Other uncontrolled, concurrent illness that would preclude study participation; or, psychiatric illness or social challenges that would entail unreasonable risk or preclude informed consent or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events

SECONDARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vonderheide, MD, DPhil, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rose S. Immunotherapy network launches first trial. Cancer Discov. 2012 Sep;2(9):760. doi: 10.1158/2159-8290.CD-ND2012-032. Epub 2012 Jul 26. No abstract available. PMID 22969103